CLINICAL TRIAL: NCT00109044
Title: Fixed Dose Comparison of Escitalopram Combination in Adult Patients With Major Depressive Disorder
Brief Title: Comparison of Escitalopram Combination in Adult Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCT-MD-35
Record Dates: First submitted 2005-04-22; First posted 2005-04-25 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder; Escitalopram
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram

INTERVENTIONS:
Drug: Escitalopram

SUMMARY:
Escitalopram is the S-enantiomer of citalopram. Both escitalopram and citalopram are selective serotonin reuptake inhibitors (SSRIs) and are used to treat depression in adults. This study is designed to evaluate the efficacy and safety of a fixed-dose escitalopram combination relative to its component monotherapies and to placebo in patients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet Diagnostic and Statistical Manual, Fourth Edition (DSM-IV) diagnostic criteria for Major Depressive Disorder.
* The patient's current depressive episode must be at least 12 weeks in duration.

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women of childbearing potential who are not practicing a reliable method of birth control.
* Patients who currently meet DSM-IV criteria for: a. bipolar disorder; b. schizophrenia or any psychotic disorder; c. obsessive-compulsive disorder; d. mental retardation or any pervasive developmental disorder or cognitive disorder.
* Patients who are considered a suicide risk.
* Patients with a history of seizure disorder, or any history of seizure, stroke, significant head injury, or any other condition that predisposes toward risk of seizure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540
Dates: Start 2005-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS)

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Southwest Health, Ltd, Phoenix, Arizona
  - Alpine Clinical Research, Boulder, Colorado
  - Radiant Research, Inc., Denver, Colorado
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Cunningham Clinical Research, LLC, Edwardsville, Illinois
  - Midwest Center for Neurobiological Medicine, Oakbrook Terrace, Illinois
  - Capital Clinical Research Associates, Rockville, Maryland
  - Summit Research Network (Michigan), Inc., Okemos, Michigan
  - CNS Research Institute, Clementon, New Jersey
  - Center for Emotional Fitness, Moorestown, New Jersey
  - Eastside Comprehensive Medical Center, New York, New York
  - Piedmont Medical Research Associates, Inc., Winston-Salem, North Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Claghorn-Lesem Research Clinic, Bellaire, Texas
  - Croft Group Research Center, San Antonio, Texas
  - Dominion Clinical Research, Midlothian, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle), LLC, Seattle, Washington